CLINICAL TRIAL: NCT04461496
Title: The Pilot Clinical Trial Comparing the Efficacy of Single-stage Multilevel Revascularization of the Iliac-femoral-popliteal Segment Using the FULL METALL JACKET Technology in Comparison With the Hybrid Revascularization Procedure
Brief Title: Full Metall Jacket Multilevel Segment
Acronym: FMJSFA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMJ
Record Dates: First submitted 2020-06-29; First posted 2020-07-08 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Superficial Femoral Artery Stenosis; Iliac Artery Occlusion
Keywords: hybrid revascularization; atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid revascularization (Active Comparator): 50 hybrid procedure
  Interventions: Procedure: Hybrid revascularization
- Full metall jacket (Experimental): 50 total endovascular interventions
  Interventions: Procedure: Full metall Jacket

INTERVENTIONS:
Procedure: Hybrid revascularization — The first stage is performed femoral-popliteal bypass surgery above the fissure of the knee joint according to conventional technology. Conduit is at the discretion of the operating surgeon. Intraoperatively bolus is administered sol. heparin 5000 IU. The second step is the puncture of the selected CFA with a retrograde installation of the introducer sheath. The iliac segment is recanalized with angioplasty and stent implantation in the affected area
  Arms: Hybrid revascularization
Procedure: Full metall Jacket — The first step is the puncture contralateral CFA with a retrograde installation of the introducer. Intraoperatively bolus is administered sol. heparin 5000 IU. A conductor is placed in the contralateral iliac artery along the conductor. A stent is implanted in the iliac artery lesion. The second stage is the recanalization of the femoral-popliteal segment with angioplasty and stent implantation in the affected area.
  Arms: Full metall jacket

SUMMARY:
Hypothesis: "Total" endovascular revascularization of a multistory lesion of the iliac-femoral-popliteal segment is safer and a better quality of life is achieved in comparison with hybrid intervention.

The lack of damage to the skin avoids complications in the postoperative and remote periods of observation, thereby improving the quality of life

DETAILED DESCRIPTION:
Mortality from cardiovascular disease occupies a leading position worldwide. Patients with atherosclerotic lesions of the peripheral arteries account for 20% of the total number of patients with cardiovascular diseases. Special attention should be paid to patients with multilevel lesions artery since the maximum reduction in blood flow leads to the development of critical limb ischemia (CLI) and a high risk of limb loss. Almost 25% of patients with CLI require multistory revascularization of the arteries of the lower extremities. In this group of patients, proximal revascularization of the only iliac segment is usually the initial approach, but in some cases leads to disappointing relief of symptoms due to concomitant severe lesions of the infra-anginal arteries. Whereas the combined implementation of femoral-popliteal bypass surgery or endovascular revascularization of SFA can increase the likelihood of ulcer healing and avoid multi-stage surgical interventions. In turn, an adequate inflow to the revascularized segment is necessary for its long-term functioning.

Femoral-popliteal bypass surgery is still the procedure of choice for long occlusions of the superficial femoral artery TASC C, D. The "total" endovascular correction (full metal jacket) may become an alternative to hybrid technology since allows for less traumatic and fully revascularization of the wall occlusal lesions of SFA. The salvation of the limb and the achievement of compensation for the clinic of chronic lower limb ischemia in patients with multi-vessel atherosclerotic lesions of the arteries of the lower extremities is possible using both hybrid procedures and endovascular reconstruction. The main goal of stenting the iliac arteries during hybrid procedures is not only to restore blood flow in the common and deep femoral arteries but also to support the long-term functioning of the femoral-popliteal shunt or stent in SFA.

Similar analogues of the comparative study of the two methods of revascularization in the world literature the investigators have not seen.

In the first group, stenting of the iliac artery under x-ray control with the bypass of the femoral-popliteal segment above the gap of the knee joint is performed. The first stage is performed femoral-popliteal bypass surgery above the fissure of the knee joint according to conventional technology. Conduit is at the discretion of the operating surgeon. Intraoperatively bolus is administered heparin 5000 IU. The second step is the puncture of the selected CFA with a retrograde installation of the introducer sheath. The iliac segment is recanalized with angioplasty and stent implantation in the affected area. In the postoperative period, clexane is administered at a prophylactic dosage of 3 days and cardiomagnyl at a dosage of 75 mg per day. Next, the patient takes dual antiplatelet therapy cardiomagnyl 75 mg + clopidogrel 75 mg for 6 months.

In the second group, stenting of the iliac artery and recanalization SFA with angioplasty and stenting under X-ray control is performed. The first step is the puncture contralateral CFA with a retrograde installation of the introducer. Intraoperatively bolus is administered heparin 5000 IU. A conductor is placed in the contralateral iliac artery along the conductor. A stent is implanted in the iliac artery lesion. The second stage is the recanalization of the femoral-popliteal segment with angioplasty and stent implantation in the affected area. In the postoperative period, a loading dose of clopidogrel 300 mg + cardiomagnyl 75 mg is taken. Next, the patient takes dual antiplatelet therapy cardiomagnyl 75 mg + clopidogrel 75 mg for 6 months.

Statistical analysis: Data processing and comparison of variables will be carried out by appropriate statistical methods with a preliminary check for compliance of the sign variability with the normal distribution, which is evaluated by the Kolmogorov-Smirnov criterion. Under the condition of the normal distribution, Student's criterion is used. A comparative assessment of qualitative characteristics is carried out using the χ2 criterion. The dynamics of the indicators in the group will be determined by the pairwise coupled option using the Student criterion with a normal distribution of indicators and using the Wilcoxon criterion - with a mismatch with the normal distribution. Comparison according to qualitative characteristics (gender, degree of ischemia, and others) will be carried out using the criteria of Pearson (Pearson) and Fisher (Fisher). In all cases, a 95% significance level is used.

ELIGIBILITY:
Inclusion Criteria:

* patients with multisegment lesions of the iliac-femoral-popliteal segment, with the distal border of the lesion above the slit of the knee joint.
* chronic ischemia 3-6 (according to Rutherford),
* the satisfactory direction of the outflow.
* Patients who gave consent to participate in this study

Exclusion Criteria:

* Chronic occlusion of the SFA at least 2cm
* Heavy calcification of SFA • Infection in the area of the access artery
* Expressed, more than 50% stenotic lesions of the infrarenal aorta
* Prolonged loss (TASC D) iliac artery on the side of revascularization
* aneurysmal widening of the infrarenal aorta and iliac arteries
* Hemodynamically significant lesions DFA
* Chronic heart failure III-IV functional class NYHA classification;
* decompensated Chronic "pulmonary" heart; • Severe hepatic or renal insufficiency (bilirubin >35 mmol/l, glomerular filtration rate <60 ml/min);
* Polyvalent drug Allergy;
* Malignant cancer in the terminal stage with a projected life span of 6 months;
* Acute stroke;
* a Pronounced calcification of the arteries of the lower limbs;
* Patients with significant lesions of the common femoral artery
* the Refusal of a patient to participate or continue to participate in the study.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2025-06-05 (Estimated); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the procedure | 24 months
  freedom from thrombosis was defined as the absence of occlusion by duplex ultrasonography or CT angiography of the treated segment
Safety of the procedure | 30 days
  bleeding according to blood loss volume (millilitres) 1. intraoperative blood loss volume; 2.Postoperative blood loss volume by duplex ultrasonography and drainage losses
Safety of the procedure | 24 months
  major adverse limb events according to clinical evaluation

SECONDARY OUTCOMES:
Primary patency | 24 months
  Primary patency rate at 24 months follow-up
Secondary patency | 24 months
  Secondary patency rate at 24 months follow-up
Changes in the patients quality of life: questionnaire | 24 months
  improving the quality of life in accordance with the questionnaire "The Short Form-36" for 24 months. The indicators of each scale are designed in such a way that the higher the value of the indicator (from 0 to 100), the better the score on the selected scale
Success of the procedure | 1 month
  the number of successful attempts
Changes in chronic lower limb ischemia at 24 months follow-up | 24 months
  Number of cases of improvement of at least 1 category of Rutherford classification for claudicants

CONTACTS AND LOCATIONS:
Locations (1):
- Meshalkin Research Institute of Pathology of Circulation, Novosibirsk, Novosibirskaya Obl, Russia